CLINICAL TRIAL: NCT06283745
Title: Randomized Clinical Trial of Intranasal Injection of Platelet-Rich Plasma for Treatment of Parosmia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Zara M. Patel, Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 73225
Record Dates: First submitted 2024-02-21; First posted 2024-02-28 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Paraosmia
MeSH Terms: conditions — Olfaction Disorders | interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: PRP injections will be given to one arm while sham saline injections will be given to the other arm.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Platelet Rich Plasma (PRP) (Active Comparator): Participants receive PRP intranasal injection into the olfactory cleft three times, separated by two weeks each. Blood is drawn from the patient. This is placed in a centrifuge and using a specialized PRP kit (Emcyte), the sequential spinning process isolates the platelet-rich plasma portion of the blood and we inject that back into the patient within the nasal cavity.
  Interventions: Other: Platelet-rich Plasma (PRP)
- Saline (Active Comparator): Participants receive saline injections into the olfactory cleft three times, separated by two weeks each. (Sham/placebo injections).
  Interventions: Other: Saline

INTERVENTIONS:
Other: Platelet-rich Plasma (PRP) — Platelet-rich plasma (PRP) intranasal injection in the treatment of qualitative olfactory dysfunction (parosmia). This is taken from a blog draw from the patient themselves, and thus no external drug/biologic product will be given - only the concentrated plasma portion from the patient's own blood.
  Arms: Platelet Rich Plasma (PRP)
Other: Saline — Saline intranasal injection (sham injection)
  Arms: Saline

SUMMARY:
This randomized clinical trial will evaluate the benefit of platelet-rich plasma (PRP) in the treatment of qualitative olfactory dysfunction (parosmia). PRP can be isolated from a patient's own blood and has been found in previous studies to have anti-inflammatory and pro-regenerative properties. It has been used across multiple specialties, such as Orthopedics, Facial Plastics, Dermatology, Neurology in injected form to treat a wide variety of tissues to encourage the body's inherent regenerative capacity. The investigators have completed a randomized controlled trial here, ending in 2022, evaluating it's use in post-SARS-CoV-2 olfactory loss which demonstrated safety and efficacy. Therefore, the investigators aim to assess the ability of PRP to improve olfactory function in patients with parosmia.

ELIGIBILITY:
Inclusion Criteria:

* Patients >= 18 years of age
* Patients who have qualitative olfactory distortion
* Etiology of qualitative olfactory distortion is due to upper respiratory infection
* Quantitative score under the 10th percentile on the SSParoT (HedRang and HedDir)
* Quantitative score ≥ 8 on the QOD.
* At least 6 months of parosmia but less than 24 months
* Patients can have been previously treated with oral and topical steroids but this is not a requirement
* Patients will receive concurrent olfactory training - the practice of smelling strong odors (standard of care)
* Be able to read and understand English
* Be able and willing to provide Informed Consent

Exclusion Criteria:

* Patients < 18 years of age, pregnant females, patients who have structural abnormalities on nasal endoscopy or radiographic imaging that would prevent injection into the olfactory cleft
* Olfactory loss due to trauma, chronic sinusitis / inflammation / polyps, neoplasms, or neurodegenerative diseases or patients who have had olfactory loss > 24 months
* Patients with bleeding disorders or on blood thinners such as coumadin and plavix

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-11-23 (Estimated); Primary Completion 2027-03-22 (Estimated); Study Completion 2027-03-22 (Estimated)

PRIMARY OUTCOMES:
Change in Sniffin Sticks Parosmia Test (SSParoT) | Assessed at baseline, 1 month, and 3 months
  The test consists of a total of 22 sticks, 11 of which are pleasant odors and 11 of which are unpleasant odors. In this test, the test subject is offered a pair of sticks, 1 with an unpleasant odor and 1 with a pleasant odor.
  The SSParoT is the first test to measure qualitative olfactory function. This test uses hedonic estimates of two oppositely odors (pleasant and unpleasant) to assess the Hedonic Range (HR) and Hedonic Direction (HD). These values represent the qualitative olfactory perception.
Change in questionnaire of olfactory disorders (QOD) scale score | Assessed at baseline, 1 month, and 3 months
  The QOD is a 25-item validated instrument in the measurement of olfactory-specific QOL (total score on 75) described by Hummel et al. Patients will undergo nasal endoscopy as part of their initial standard of care appointment to exclude structural causes of smell loss including mass or tumor, as well as ensuring there is no structural obstruction to the olfactory cleft such as severe septal deviation.

CONTACTS AND LOCATIONS:
Overall Officials: Zara Patel, MD, Principal Investigator — Stanford Otolaryngology - Head and Neck Surgery
Locations (1):
- Stanford Sinus Center / Stanford University School of Medicine, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Prognosis and persistence of smell and taste dysfunction in patients with covid-19: meta-analysis with parametric cure modelling of recovery curves. BMJ. 2022 Aug 9;378:o1939. doi: 10.1136/bmj.o1939. No abstract available. PMID 35944915
- [Background] Pence TS, Reiter ER, DiNardo LJ, Costanzo RM. Risk factors for hazardous events in olfactory-impaired patients. JAMA Otolaryngol Head Neck Surg. 2014 Oct;140(10):951-5. doi: 10.1001/jamaoto.2014.1675. PMID 25170573
- [Background] Pellegrino R, Mainland JD, Kelly CE, Parker JK, Hummel T. Prevalence and correlates of parosmia and phantosmia among smell disorders. Chem Senses. 2021 Jan 1;46:bjab046. doi: 10.1093/chemse/bjab046. PMID 34698820
- [Background] Chang MT, Patel ZM. Novel Therapies in Olfactory Disorders. Curr Otorhinolaryngol Rep. 2022;10(4):427-432. doi: 10.1007/s40136-022-00436-z. Epub 2022 Oct 22. PMID 36312744
- [Background] Yan CH, Mundy DC, Patel ZM. The use of platelet-rich plasma in treatment of olfactory dysfunction: A pilot study. Laryngoscope Investig Otolaryngol. 2020 Feb 21;5(2):187-193. doi: 10.1002/lio2.357. eCollection 2020 Apr. PMID 32337347
- [Background] Zahn J, Loibl M, Sprecher C, Nerlich M, Alini M, Verrier S, Herrmann M. Platelet-Rich Plasma as an Autologous and Proangiogenic Cell Delivery System. Mediators Inflamm. 2017;2017:1075975. doi: 10.1155/2017/1075975. Epub 2017 Aug 6. PMID 28845088
- [Background] Kaux JF, Croisier JL, Forthomme B, Le Goff C, Buhler F, Savanier B, Delcour S, Gothot A, Crielaard JM. Using platelet-rich plasma to treat jumper's knees: Exploring the effect of a second closely-timed infiltration. J Sci Med Sport. 2016 Mar;19(3):200-204. doi: 10.1016/j.jsams.2015.03.006. Epub 2015 Mar 21. PMID 25840691
- [Background] Chen SR, Shen YP, Ho TY, Li TY, Su YC, Chou YC, Chen LC, Wu YT. One-Year Efficacy of Platelet-Rich Plasma for Moderate-to-Severe Carpal Tunnel Syndrome: A Prospective, Randomized, Double-Blind, Controlled Trial. Arch Phys Med Rehabil. 2021 May;102(5):951-958. doi: 10.1016/j.apmr.2020.12.025. Epub 2021 Feb 3. PMID 33548206
- [Background] Anjayani S, Wirohadidjojo YW, Adam AM, Suwandi D, Seweng A, Amiruddin MD. Sensory improvement of leprosy peripheral neuropathy in patients treated with perineural injection of platelet-rich plasma. Int J Dermatol. 2014 Jan;53(1):109-13. doi: 10.1111/ijd.12162. Epub 2013 Oct 29. PMID 24168291
- [Background] Hibner M, Castellanos ME, Drachman D, Balducci J. Repeat operation for treatment of persistent pudendal nerve entrapment after pudendal neurolysis. J Minim Invasive Gynecol. 2012 May-Jun;19(3):325-30. doi: 10.1016/j.jmig.2011.12.022. Epub 2012 Feb 4. PMID 22305742
- [Background] Yan CH, Jang SS, Lin HC, Ma Y, Khanwalkar AR, Thai A, Patel ZM. Use of platelet-rich plasma for COVID-19-related olfactory loss: a randomized controlled trial. Int Forum Allergy Rhinol. 2023 Jun;13(6):989-997. doi: 10.1002/alr.23116. Epub 2022 Dec 21. PMID 36507615
- [Background] Liu DT, Welge-Lussen A, Besser G, Mueller CA, Renner B. Assessment of odor hedonic perception: the Sniffin' sticks parosmia test (SSParoT). Sci Rep. 2020 Oct 22;10(1):18019. doi: 10.1038/s41598-020-74967-0. PMID 33093474
- [Background] Frasnelli J, Hummel T. Olfactory dysfunction and daily life. Eur Arch Otorhinolaryngol. 2005 Mar;262(3):231-5. doi: 10.1007/s00405-004-0796-y. Epub 2004 May 5. PMID 15133691